CLINICAL TRIAL: NCT00554918
Title: A Randomised Phase II Feasibility Study of Docetaxel (Taxotere®) Plus Prednisolone vs. Docetaxel (Taxotere®) Plus Prednisolone Plus Zoledronic Acid (Zometa®) vs. Docetaxel (Taxotere®) Plus Prednisolone Plus Strontium-89 vs. Docetaxel (Taxotere®) Plus Prednisolone Plus Zoledronic Acid (Zometa®) Plus Strontium-89 in Hormone Refractory Prostate Cancer Metastatic to Bone.
Brief Title: Docetaxel and Prednisolone With or Without Zoledronic Acid and/or Strontium Chloride Sr 89 in Treating Patients With Prostate Cancer Metastatic to Bone That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CRUK-TRAPEZE-2100; CDR0000574585 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2004-002295-41; EU-20782; ISRCTN12808747; SANOFI-AVENTIS-CRUK-TRAPEZE-21; NOVARTIS-CRUK-TRAPEZE-2100
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-04

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Docetaxel; Prednisolone; Zoledronic Acid; strontium chloride

INTERVENTIONS:
Drug: docetaxel
Drug: prednisolone
Drug: zoledronic acid
Procedure: quality-of-life assessment
Radiation: strontium chloride Sr 89

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisolone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Zoledronic acid may help relieve some of the symptoms caused by bone metastases. Radioactive substances, such as strontium chloride Sr 89, may help relieve bone pain caused by prostate cancer. Giving docetaxel together with prednisolone with or without zoledronic acid and/or strontium chloride Sr 89 may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying the side effects and how well giving docetaxel together with prednisolone works with or without zoledronic acid and/or strontium chloride Sr 89 in treating patients with prostate cancer metastatic to bone that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the toxicity and tolerability of docetaxel with zoledronic acid.
* To assess the toxicity and tolerability of docetaxel with strontium chloride Sr 89.
* To assess the toxicity and tolerability of docetaxel with zoledronic acid and strontium chloride Sr 89.

Secondary

* Compare health economic endpoints between the treatment groups.
* Compare changes in bone mineral density between the treatment groups.
* Compare the biological profiling for prognostic and predictive indicators between the treatment groups.

Tertiary

* Compare median time to disease progression between the treatment groups.
* Compare pain progression-free survival (PFS) between the treatment groups.
* Compare PSA PFS between the treatment groups.
* Compare pain response between the treatment groups.
* Compare overall survival between the treatment groups.
* Compare quality of life between the treatment groups.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment center and ECOG performance status (0 vs 1 vs 2). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive docetaxel IV on day 1 and oral prednisolone once daily.
* Arm II: Patients receive docetaxel and prednisolone as in arm I and zoledronic acid IV over 15 minutes on day 1.
* Arm III: Patients receive docetaxel and prednisolone as in arm I and a single dose of strontium chloride Sr 89 IV on day 7 of course 2.
* Arm IV: Patients receive docetaxel and prednisolone as in arm I, zoledronic acid as in arm II, and strontium chloride Sr 89 as in arm III.

Treatment with docetaxel, prednisolone, and zoledronic acid repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Strontium chloride Sr 89 is given as a one time single dose.

Quality of life is assessed using the Euroqual (EQ-5D) and FACT-P at baseline and every 3 months during follow up.

After completion of study, patients are followed every 3 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or cytologically proven prostate adenocarcinoma
  * Multiple sclerotic bone metastases with PSA ≥ 100 ng/mL without histological confirmation
* Radiological evidence of bone metastasis
* Prior hormonal therapy for prostate cancer including ≥ 1 of the following:

  * Bilateral orchidectomy
  * Medical castration by luteinizing hormone-releasing hormone (LHRH) agonist therapy

    * If receiving LHRH agonist therapy alone, this therapy should be continued
* Documented disease progression, defined by one of the following:

  * Progressive disease after discontinuing hormone therapy
  * Elevated and rising PSA, defined as 2 consecutive increases in PSA documented over a previous reference value
  * PSA > 5ng/mL
  * Progression of any unidimensionally or bidimensionally measurable malignant lesion
  * At least 1 new lesion identified on bone scan
* No known brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Hemoglobin ≥ 10g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 1.5 times ULN (unless related to hepatic metastatic disease, where patients may be entered after discussion with one of the clinical advisors)
* Serum bilirubin ≤ 1.5 times ULN
* Physically fit enough to receive trial treatment
* No malignant disease within the past 5 years, other than adequately treated basal cell carcinoma
* No symptomatic peripheral neuropathy ≥ grade 2 (NCI CTC)
* No known hypersensitivity to bisphosphonates
* No condition, in the opinion of the investigator, that may interfere with the safety of the patient or evaluation of the study objectives

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior flutamide, nilutamide, or cyproterone acetate with evidence of disease progression since cessation
* At least 6 weeks since prior bicalutamide with evidence of disease progression since cessation
* At least 4 weeks since prior estramustine and any adverse events must have resolved
* At least 2 months since prior treatment with a bisphosphonate for any reason
* No treatment with any other investigational compound within the past 30 days
* No prior cytotoxic chemotherapy for hormone refractory prostate cancer (HRPC), other than estramustine monotherapy
* No prior radionuclide therapy for HRPC
* No prior radiotherapy to more than 25% of the bone marrow or whole pelvic irradiation
* No concurrent enrollment in any other investigational clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety
Toxicity and tolerability of docetaxel and zoledronic acid
Toxicity and tolerability of docetaxel and strontium chloride Sr 89
Toxicity and tolerability of docetaxel, zoledronic acid, and strontium chloride Sr 89

SECONDARY OUTCOMES:
Health Care economic analysis
Changes in bone mineral density
Median time to disease progression
Pain progression-free survival (PFS)
PSA PFS
Pain response
Overall survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D. James, MD, Study Chair — University Hospital Birmingham
Locations (16):
- United Kingdom (16):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Ipswich Hospital, Ipswich, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Royal Marsden - Surrey, Sutton, England
  - Walsall Manor Hospital, Walsall, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales

REFERENCES:
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906